CLINICAL TRIAL: NCT03162133
Title: Evaluating the Impact of Baduanjin Exercise Intervention on Quality of Life in Breast Cancer Survivors Receiving Aromatase Inhibitor Therapy：: A Pilot Study
Brief Title: Evaluating the Impact of Baduanjin Exercise Intervention on Quality of Life in Breast Cancer Survivors Receiving Aromatase Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Guangzhou Sport University (Other)
Responsible Party: Principal Investigator, KunWang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20170217
Record Dates: First submitted 2017-05-12; First posted 2017-05-22 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Survivors Receiving Aromatase Inhibitor Therapy
Keywords: Breast Cancer; Aromatase Inhibitor Therapy; Baduanjin Exercise
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): After completing the baseline tests, participants in exercise group were instructed to attend 90-minute, supervised Baduanjin exercise 2 times per week. The Baduanjin intervention used the standardized Baduanjin training program, designed by the General Administration of Sports of China. Two senior Baduanjin teachers from Guangzhou Sports University conducted the training.
  Interventions: Other: Baduanjin exercise
- Waiting list Control group (Experimental): Participants assigned to the wait-list control were told to continue performing their usual care and daily activities, and to refrain from doing any Baduanjin exercise.
  After their post-assessment they were able to attend the Baduanjin classes.
  Interventions: Other: Baduanjin exercise

INTERVENTIONS:
Other: Baduanjin exercise

SUMMARY:
A 12-week randomized controlled trail was conducted in 72 Chinese breast cancer survivors who had received aromatase inhibitors treatment for more than 6 months. All participants were assigned to either 12 weeks of Baduanjin classes which involved to two 90-minute sessions per week or a wait-list control. Participants completed fitness assessments, measurements of lipopolysaccharide-stimulated production of proinﬂammatory cytokines interleukin-6 (IL-6), tumor necrosis factor alpha (TNF-α), interleukin-1β(IL-1β) ,C-reactive protein (CRP) ，BMI，BMD and questionnaires to measure QoL, fatigue, sleep quality, Aromatase Inhibitor-Induced Arthralgia, symptoms of climacteric syndrome were completed at baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed as stage I to III breast cancer 0.5 to 4.0 years before enrollment
* Taking an AI (aromatase inhibitors )，and had been receiving an AI for at least 6 months

Exclusion Criteria:

* A prior history of breast or any other cancer except basal or squamous cell skin cancer Inﬂammatory breast cancer
* With exercise contraindications：chronic obstructive pulmonary disease, uncontrolled hypertension, evidence of liver or kidney failure, symptomatic ischemic heart disease ,conditions involving the immune system such as autoimmune and/or inﬂammatory diseases, cognitive impairment, alcohol/drug abuse
* Current Baduanjin practice (within the last 6 months), and/or previous Baduanjin practice for more than 3 months
* Women reporting 5 hours or more of vigorous physical activity per week

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quality of Life (QoL) at 3 months | at baseline and 3 months
  European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 version 3 (EORTC QLQ-C30)

SECONDARY OUTCOMES:
Change from Baseline IL-6 at 3 months | at baseline and 3 months
  proinﬂammatory cytokines interleukin-6
Change from Baseline Fatigue at 3 months | at baseline and 3 months
  Piper fatigue questionnaire
Change from Baseline sleep quality at 3 months | at baseline and 3 months
  Pittsburgh sleep quality index, PSQI
Change from Baseline Aromatase Inhibitor-Induced Arthralgia at 3 months | at baseline and 3 months
  Brief Pain Inventory-Short Form
Change from Baseline Symptoms of climacteric syndrome at 3 months | at baseline and 3 months
  Kupperman Index
Change from Baseline BMD at 3 months | at baseline and 3 months
  Bone mineral density
Change from Baseline BMI at 3 months | at baseline and 3 months
  Body Mass Index
Change from Baseline Aerobic Fitness Assessment at 3 months | at baseline and 3 months
  Six-min walk test (6MWT)
Change from Baseline Muscle strength test at 3 months | at baseline and 3 months
  Upper strength: hand grip (measured by a dynamometer; the average of 3 readings) lower limb strength：sit-to-stand (measured as number of reps in a 30-s period)
Change from Baseline Flexibility test at 3 months | at baseline and 3 months
  Test of scratching his back and Sit in the chair and reach
Change from Baseline Balance test at 3 months | at baseline and 3 months
  stand on one foot
Change from Baseline TNF-α at 3 months | at baseline and 3 months
  tumor necrosis factor alpha
Change from Baseline IL-1β at 3 months | at baseline and 3 months
  interleukin-1β
Change from Baseline CRP at 3 months | at baseline and 3 months
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided